CLINICAL TRIAL: NCT00113282
Title: Study of the Immunological Efficacy of Adding Subcutaneous Interleukin-2 (IL-2) to an Optimized Antiretroviral Regimen in HIV-1-infected Subjects Experiencing Therapeutic Failure on an Ongoing Antiretroviral Combination With a CD4 Cell Count ≤ 200/mm3 ANRS 123 Trial
Brief Title: Efficacy of Adding Interleukin-2 to an Optimized Antiretroviral Regimen in HIV Patients in Therapeutic Failure (ANRS123)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Chiron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-001329-29; ANRS123
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2009-06

CONDITIONS: HIV Infections
Keywords: Treatment failure; Acquired Immunodeficiency Syndrome; Interleukin-2; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Interleukin-2 (IL-2)

SUMMARY:
Interleukin-2 (IL-2) increases the number of CD4 cells in HIV-1 infected patients with a CD4 cell count over 200/mm3, but its activity in patients with treatment failure and low CD4 cell counts is unknown. This study will test the efficacy and safety of IL-2 with an optimized antiretroviral regimen in patients with a CD4 count below 200/mm3 and a plasma viral load above 10,000 HIV RNA copies/ml.

DETAILED DESCRIPTION:
IL-2 is produced naturally in the body and helps CD4 cells multiply. In earlier studies in HIV-infection, most of the patients with a controlled viral load and a high level of CD4 count (over 200/mm3) who received IL-2, experienced an increase of their CD4 cell count superior to what is observed with antiretroviral therapy alone.

The efficacy of IL-2 when the viral load is high and the CD4 cell count is low is not known. The purpose of this multicentric national study is to compare the effects of an optimized antiretroviral regimen with or without IL-2.The choice of the antiretroviral regimen will be made from a genotype resistance test.

Ninety eight HIV-1-infected patients experiencing advanced treatment failure with a CD4 count below 200/mm3 and a plasma viral load above 10,000 HIV RNA copies/ml, will be randomly assigned to one of two treatment groups: with or without IL-2.

The group with IL-2 will receive a dose of 4.5 million International units by subcutaneous injection twice a day for 5 days (up to a total of 8 cycles, ending at Week 42), the first two cycles 4 weeks apart, the following cycles 6 weeks apart.

Evaluation will be done at week 52 and further at W76. The primary endpoint is the proportion of patients reaching an absolute CD4 count over 200/mm3 at Week 52. Secondary endpoints include the proportion of patients increasing their CD4 count over 50/mm3 between Week 00 and Week 24,and between Week 00 and Week 52, the occurrence of HIV-related events, drug safety and the evolution of CD4 cells and of HIV RNA and HIV DNA loads over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with proven HIV-1-infection
* Prior or current exposition to at least 1 molecule from each of the 3 antiretroviral classes (NRTI, NNRTI and PI)
* In a situation of therapeutic failure on an ongoing regimen

Exclusion Criteria:

* Patients included in the Macrolin® expanded French access program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-06; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
proportion of patients reaching an absolute CD4 count over 200/mm3 at Week 52 (W52)

SECONDARY OUTCOMES:
group B or C events (1993 CDC classification of HIV infection)between Week 00 and Week 96
median value of the CD4 count at W52
evolution of the CD4 count during the study
time to the first visit with a CD4 count ≥ 200/mm3
tolerance of IL-2
tolerance of antiretroviral drugs
evolution of the plasma HIV RNA load at W64 and W76
evolution of the HIV DNA level in PBMCs at W64 and W76
number of modifications of antiretroviral regimen until W52
clinical status at W64 and W76
CD4 count at W64, W76 and W96
plasma HIV RNA load at W64, W76 and W96
number of modifications of antiretroviral regimen at W64 and W76
proportion of patients increasing their CD4 count over 50/mm3 between Week 00 and Week 24, and between Week 00 and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Chêne, Pr, Study Chair — Inserm Unite 593; Jean Paul VIARD, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker service des Maladies Infectieuses, Paris, France